CLINICAL TRIAL: NCT03156933
Title: Alternative Splicing and Leukemia Initiating Cells
Acronym: ASLIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0800
Record Dates: First submitted 2017-04-04; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Splicing variants: Sample of acute myeloid leukaemia primary cells
  Interventions: Other: Assessment of splicing variants

INTERVENTIONS:
Other: Assessment of splicing variants — This is a biological study with primary samples without any intervention on patients.

SUMMARY:
Aberrant RNA splicing and mutations in spliceosome complex in acute myeloid leukaemia (AML) are frequent. It have been shown that some splicing variants had a prognostic value in AML.

AML are characterized by their propensity to relapse because of the persistence of leukaemia initiating cells (LICs).

The aim of this study is to determine the splice variants on AML initiator cells and define a splicing pattern.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old
* Patients treated at the south lyon hospital center
* Patients with a diagnosis of acute myeloid leukemia confirmed in cytology and whose involvement of the 11q23 locus was confirmed by in situ hybridization
* Patients for whom a sample is available in the cytogenetic laboratory of the south lyon hospital center

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 11q23 acute myeloid leukaemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Polymerase chain reaction | 1 month
  Transcriptome analysis to determine the splicing variants on acute myeloid leukaemia initiator cells.
  The analysis will focus on the gene encoding ABCA3 transporter and genes known to be mutated in patients with acute myeloid leukemia (FLT3, NPM1, c-Kit, N et K-RAS).
  The duration of selection of samples is estimated to be one month.
Ribonucleic acid sequencing | 1 month
  Transcriptome analysis to determine the splicing variants on acute myeloid leukaemia initiator cells.
  The analysis will focus on the gene encoding ABCA3 transporter and genes known to be mutated in patients with acute myeloid leukemia (FLT3, NPM1, c-Kit, N et K-RAS).
  The duration of selection of samples is estimated to be one month.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne PAUBELLE, MD, PhD, Principal Investigator — Service d'hématologie du Centre Hospitalier Lyon Sud
Locations (1):
- Service d'hématologie du Centre Hospitalier Lyon Sud, Pierre-Bénite, France